CLINICAL TRIAL: NCT06959797
Title: Randomized Cross-over Study Comparing Insulin Pump Versus Full Closed-loop Automated Insulin Therapy in Type 2 Diabetic Patients Previously Treated With Insulin Pumps
Brief Title: Insulin Pump Versus Full Closed-loop for Type 2 Diabetes
Acronym: IA-DT2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Abbott (Industry); mylife Diabetes Care AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23-0251; ID RCB 2023-A02593-42 (Other: ANSM)
Record Dates: First submitted 2025-04-24; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes, automated insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Clinical Investigation of a Medical Device (IC-DM)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Closed loop then Open loop) (Experimental): Ypsomed pump (Ypsomed), CamAPS HX application activated, Android smartphone. Freestyle 3 sensors (Abbott) Then Ypsomed pump (Ypsomed). Android smartphone. Freestyle 3 sensors (Abbott)
  Interventions: Device: Closed loop; Device: Open loop
- Arm II (Loop Open then Loop Closed) (Experimental): Ypsomed pump (Ypsomed). Android smartphone. Freestyle 3 sensors (Abbott) Then Ypsomed pump (Ypsomed), CamAPS HX application activated, Android smartphone. Freestyle 3 sensors (Abbott)
  Interventions: Device: Closed loop; Device: Open loop

INTERVENTIONS:
Device: Closed loop — Ypsomed pump (Ypsomed), CamAPS HX application activated, Android smartphone. Freestyle 3 sensors (Abbott)
Device: Open loop — Ypsomed pump (Ypsomed). Android smartphone. Freestyle 3 sensors (Abbott)

SUMMARY:
The aim of the study is to compare, in a population of patients with type 2 diabetes, open-loop insulin pump treatment with the CamAPS HX (Camdiab) Fully Closed Loop Automated Insulin Therapy system, on the efficacy and safety of use of the Fully Closed Loop, as well as on psycho-social criteria of device acceptability, quality of life and diabetes burden. This is an open, multi-center, randomized, cross-over study, based on several observational or controlled trials carried out in Cambridge by Prof. Hovorka's team (see paragraph 4 below). The study will comprise a run-in phase followed by a 1st sequence in which randomized patients will use the Ypsomed pump (Ypsomed) and the FreeStyle Libre 3 sensor in open loop for 12 weeks Versus the Ypsomed pump (Ypsomed) coupled with the CamAPS HX algorithm and the FreeStyle Libre 3 sensor in full closed loop. At the end of this 1ère sequence, all patients will undergo a 2-4 week washout, during which they will use the Ypsomed pump and the FreeStyle Libre 3 sensor in open loop, and then in the 2nd sequence of the study, patients will switch to the other treatment for a further 12 weeks. A total of 80 patients on insulin pumps for at least 6 months will be recruited from 9 French centers. All patients will receive training in the use of the Ypsomed pump, the FreeStyle Libre 3 sensor and the CamAPS HX algorithm. The primary objective is Time on Target 70-180 mg/dl of 24h measured during the 12 weeks of each therapeutic period. Secondary objectives will be Time in Target 70-180 mg/dl day and night, Time above Target > 180 mg/dl and > 250 mg/dl, Time below Target < 70 mg/dl and < 54 mg/dl, time in the narrow target range 70-140 mg/dL, mean 24h blood glucose and glycemic variability measured over the 12 weeks of each treatment sequence, HbA1c, weight, total insulin dose and psychosocial endpoints assessed at the start and end of each treatment sequence. Safety data studied will include diabetes-related adverse events (ketoacidosis, symptomatic and severe hypoglycemia) and medical device-related adverse events (pump and sensor).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Type 2 diabetes for at least 12 months
* On insulin pump for at least 6 months, without/with adjuvant treatment exclusively with GLP1-Ra, iSGLT2, metformin for at least 3 months
* Autonomy in the management of the pump and the glucose sensor
* HbA1c ≥ 7.5% and < 12
* Participant's agreement to wear and use the Ypsomed with the CamAPS HX algorithm and Free Style Libre 3 sensor, and to honor the study visit schedule
* For women of childbearing age, effective contraception is required (estrogen-progestin pill, IUD, implant).

Exclusion Criteria:

* Type 1 diabetes or monogenic diabetes
* Use of U500 or U200 insulin concentrate in the pump in the last 3 months
* Allergy to insulin or to the adhesives used
* Severe insulin resistance defined by a daily insulin requirement of more than 1.5 U/kg
* History of severe hypoglycemia > 1 time in the last 6 months.
* Current or planned use of steroids (oral, injectable) or any treatment likely to have an impact on blood glucose levels within the last 30 days.
* Current or planned pregnancy, breastfeeding
* Severe renal failure defined as GFR < 30 ml/mn
* Proliferative retinopathy or severe maculopathy with risk of worsening during the study
* Vision or hearing problems that could compromise safe use of the device
* Acute vascular event within the last 3 months
* No autonomy for pump treatment
* Alcohol or substance abuse
* Legal protection (guardianship, curatorship)
* Any somatic or psychological condition compromising participation in the study
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Time on target [70-180] mg/dl over 24h for the 12 weeks of each treatment sequence | from baseline for the 12 weeks of each treatment sequence
  Time on target [70-180] mg/dl over 24h for the 12 weeks of each treatment sequence

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France